CLINICAL TRIAL: NCT02068170
Title: Risk of QT-prolongation and Torsade de Pointes in Patients Treated With Acute Medication in a University Hospital
Acronym: RISQ-PATH
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Eline Vandael, PhD-student, KU Leuven
Other Study IDs: EV003
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Delirium; QT-prolongation
Keywords: QT-prolongation; Torsade de Pointes; QT-prolonging drugs
MeSH Terms: conditions — Delirium; Long QT Syndrome; Torsades de Pointes | interventions — Haloperidol; Erythromycin; Trimethoprim, Sulfamethoxazole Drug Combination; Methadone; Tacrolimus; Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 1 blood sample (plasma) to measure the blood concentration of the drug
  * 1 blood sample (DNA) to store in a biobank for additional research
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients treated with a potentional QT-prolonging drug
  Interventions: Drug: Haloperidol, azi/clari/erythromycin, levo/moxifloxacin, co-trimoxazole, vori/keto/flu/itraconazole, methadone, tacrolimus, sunitinib

INTERVENTIONS:
Drug: Haloperidol, azi/clari/erythromycin, levo/moxifloxacin, co-trimoxazole, vori/keto/flu/itraconazole, methadone, tacrolimus, sunitinib
  Other Names: haloperidol: Haldol, ATC-code: N05AD01; azithromycin: Zitromax, ATC-code: J01FA10; clarithromycin: Biclar, ATC-code: J01FA09; erythromycin: Erytroforte, ATC-code: J01FA01; levofloxacin: Tavanic, ATC-code: J01MA12; moxifloxacin: Avelox, ATC-code: J01MA14; co-trimoxazole: Bactrim, Eusaprim, ATC-code: J01EE01; voriconazole: Vfend, ATC-code: J02AC03; ketoconazole: Nizoral, ATC-code: J02AB02; fluconazole: Diflucan, ATC-code: J02AC01; itraconazole: Sporanox, ATC-code: J02AC02; methadone: ATC-code: N07BC02; tacrolimus: Prograft, Advagraft, ATC-code: L04AD02; sunitinib: Sutent, ATC-code: L01XE04

SUMMARY:
A prospective, observational study in a university hospital (UZ Leuven). Patients are included when they are treated with a potentional QT-prolonging drug: haloperidol for delirium, antibiotics (moxifloxacin, levofloxacin, azithromycin, clarithromycin, erythromycin, co-trimoxazole), antimycotics (ketoconazole, itraconazole, fluconazole, voriconazole), methadone, tacrolimus and oral oncolytics.

An ECG is taken before the administration of the drug and 3-5 days after starting the drug to investigate the change in duration of the QTc-interval. Risk factors for developing QT-prolongation will be documented. Together with ECG2, an additional blood sample will be collected to measure the blood concentration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* treatment with a potentional QT-prolonging drug of our list
* inpatient of UZ Leuven, admitted on one of the participating wards

Exclusion Criteria:

* < 18 years old
* DNR-code 3
* not possible to take an ECG before the start of haloperidol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with acute potentional QT-prolonging medication. In a university hospital.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change in QTc-interval (corrected for heart rate) | before and 3-5 days after the start of a potentional QT-prolonging drug

CONTACTS AND LOCATIONS:
Overall Officials: Eline Vandael, PhD-student, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Vandael E, Vandenberk B, Vandenberghe J, Spriet I, Willems R, Foulon V. Development of a risk score for QTc-prolongation: the RISQ-PATH study. Int J Clin Pharm. 2017 Apr;39(2):424-432. doi: 10.1007/s11096-017-0446-2. Epub 2017 Mar 9. PMID 28281228